CLINICAL TRIAL: NCT00039195
Title: Risk-Adapted Therapy for Patients With Untreated Age-Adjusted International Prognostic Index II or III Diffuse Large B Cell Lymphoma
Brief Title: Chemotherapy and Rituximab With or Without Total-Body Irradiation and Peripheral Stem Cell Transplant in Treating Patients With Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Bristol-Myers Squibb (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-142; MSKCC-01142; NCI-G02-2069
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Results first posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-06

CONDITIONS: Lymphoma
Keywords: stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Filgrastim; Rituximab; Carboplatin; Cyclophosphamide; Doxorubicin; Etoposide; Ifosfamide; Prednisone; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

ARMS (1):
- Induction R-CHOPac Therapy for patients with B-Cell Lymphoma (Experimental): Patients received 4 cycles if accelerated R-CHOP (cyclophosphamide. doxorubicin, vincristine and prednisone + rituximab) followed by 3 cycles ICE (ifosfamide, carboplatin and etoposide) consolidation therapy.
  Interventions: Biological: filgrastim; Biological: rituximab; Drug: carboplatin; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: prednisone; Drug: vincristine sulfate; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
Biological: rituximab
Drug: carboplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Drug: prednisone
Drug: vincristine sulfate
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Combining chemotherapy with monoclonal antibody therapy, total-body irradiation, and peripheral stem cell transplant may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving chemotherapy with rituximab followed by combination chemotherapy with or without rituximab, total-body irradiation, and peripheral stem cell transplant works in treating patients with lymphoma.

DETAILED DESCRIPTION:
OUTLINE: Patients are stratified according to risk (low-intermediate vs high-intermediate or high).

Patients receive induction chemotherapy comprising cyclophosphamide IV, doxorubicin IV over 15 minutes, and vincristine IV over 1-2 minutes on day 1; oral prednisone once daily on days 1-5; and filgrastim (G-CSF) subcutaneously (SC) once daily on days 7-11 or PEG-filgrastim once at least 24 hours after infusion. Patients also receive rituximab IV 2-3 days apart for a total of 2 doses during the week prior to the first course of chemotherapy and on day 1 of courses 2-4 of chemotherapy. Treatment repeats every 14 days for a total of 4 courses in the absence of disease progression or unacceptable toxicity.

After the completion of induction chemotherapy, patients undergo CT scan and positron emission tomography (PET) scanning. If the PET scan is positive in one or more nodal sites, a repeat biopsy is performed. Patients with a negative PET scan OR a negative repeat biopsy (including no evidence of lymphoma on repeat bone marrow biopsy) are assigned to receive regimen A for consolidation therapy. Patients with a positive repeat biopsy are assigned to receive regimen B for consolidation therapy.

* Regimen A: Patients receive consolidation chemotherapy comprising etoposide IV over 1 hour on days 1-3, ifosfamide IV continuously over 24 hours on day 2, carboplatin IV on day 2, and G-CSF SC once daily on days 5-12 or PEG-filgrastim once at least 24 hours after infusion. Treatment repeats every 14 days for a total of 3 courses in the absence of disease progression or unacceptable toxicity.
* Regimen B: Patients receive consolidation chemotherapy as in regimen A for 3 courses. Patients also receive rituximab IV on days -3 to -1 of course 3 of chemotherapy. Patients undergo leukapheresis at the completion of course 3 (G-CSF continues from day 5 until the end of leukapheresis). After completion of leukapheresis, patients begin a regimen of high-dose chemoradiotherapy comprising either total body irradiation twice daily on days -10 to -7 and ifosfamide IV over 1 hour and etoposide IV continuously on days -6 to -2 or BEAM chemotherapy comprising carmustine, etoposide, cytarabine, and melphalan. Autologous peripheral blood stem cells (APBSC) are reinfused on day 0. Patients also receive G-CSF SC daily beginning on day 5 and continuing until blood counts recover. Beginning on day 42 post-APBSC, if blood counts have recovered, patients receive rituximab IV once weekly for 4 weeks. Rituximab is repeated beginning on day 180 in the absence of disease progression.

Patients who receive consolidation therapy on regimen A are followed at 4-6 weeks after chemotherapy and patients who receive consolidation therapy on regimen B are followed at 90-120 days after transplantation. All patients are followed closely for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 40-98 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed aggressive diffuse large B-cell lymphoma
* CD20-positive disease
* Age-adjusted International Prognostic Index II or III defined by the presence of at least 1 of the following:

  * Karnofsky performance status 10-70%
  * Lactate dehydrogenase greater than 200 U/L
  * Stage III or IV disease
* Positron emission tomography avid measurable disease
* No CNS involvement

PATIENT CHARACTERISTICS:

Age:

* 18 to 64

Performance status:

* See Disease Characteristics

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count greater than 50,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL unless history of Gilbert's disease or pattern consistent with Gilbert's disease
* Hepatitis B surface antigen and hepatitis C antibody negative
* No chronic, active, or persistent hepatitis

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min
* No chronic renal insufficiency

Cardiovascular:

* Ejection fraction at least 50% by echocardiogram or MUGA scan
* No myocardial infarction within the past 6 months
* No unstable angina
* No cardiac arrhythmias except chronic atrial fibrillation

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* HIV negative
* No other medical illness that would preclude study
* No uncontrolled infection
* No other malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy for malignancy

Chemotherapy:

* No prior chemotherapy for malignancy

Endocrine therapy:

* Prior steroids allowed if received no more than 1 week of therapy

Radiotherapy:

* No prior radiotherapy for malignancy

Surgery:

* No prior surgery for malignancy

Other:

* No other prior therapy for malignancy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2006-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Moskowitz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Bantilan KS, Smith AN, Maurer MJ, Teruya-Feldstein J, Matasar MJ, Moskowitz AJ, Straus DJ, Noy A, Palomba ML, Horwitz SM, Hamlin PA, Portlock CS, Cerhan JR, Habermann TM, Salles GA, Nowakowski GS, Moskowitz CH, Zelenetz AD. Matched control analysis suggests that R-CHOP followed by (R)-ICE may improve outcome in non-GCB DLBCL compared with R-CHOP. Blood Adv. 2024 May 14;8(9):2172-2181. doi: 10.1182/bloodadvances.2023011408. PMID 38271621

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction R-CHOPac Therapy: Induction R-CHOPac Therapy for patients with B-Cell Lymphoma
Period: Overall Study
Arm/Group | Induction R-CHOPac Therapy
Started | 98
Completed | 98
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Induction R-CHOPac Therapy
Number analyzed (Participants) | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 97
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 56
Region of Enrollment [Number; unit: participants]
  United States | 98

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Kaplan-Meier estimates will be used to verify the progression free survival.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients progression free
Arm/Group | Induction R-CHOPac Therapy
Number analyzed (Participants) | 98
percentage of patients progression free | 79 [69 to 89]

ADVERSE EVENTS:
Arm/Group | Induction R-CHOPac Therapy
Serious Adverse Events (participants affected / at risk) | 20/98
Other Adverse Events (participants affected / at risk) | 98/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction R-CHOPac Therapy (N=98)
Abdominal pain/cramping (Gastrointestinal disorders) | 1 (1)
Arachnoiditis (Musculoskeletal and connective tissue disorders) | 1 (1)
Constitutional symptoms, other (General disorders) | 1 (1)
Delusions (Nervous system disorders) | 1 (1)
Febrile neutropenia (General disorders) | 8 (8)
Fever (General disorders) | 1 (1)
GI, other (Gastrointestinal disorders) | 2 (2)
Headache (General disorders) | 1 (1)
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage, other (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Cardiac disorders) | 2 (2)
Ileus (or neuroconstipation) (Gastrointestinal disorders) | 1 (1)
Infection without neutropenia (Infections and infestations) | 3 (3)
Radiation mucositis (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neuropathy-sensory (Nervous system disorders) | 1 (1)
Neutrophils (Blood and lymphatic system disorders) | 2 (2)
Pain - Stomach (Gastrointestinal disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 2 (2)
Pulmonary, other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Supravent arrhythmia (Cardiac disorders) | 1 (1)
Syncope (General disorders) | 1 (1)
Thrombosis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction R-CHOPac Therapy (N=98)
Alkaline phosphatase (Metabolism and nutrition disorders) | 8 (8)
Bilirubin (Metabolism and nutrition disorders) | 20 (20)
Creatinine (Metabolism and nutrition disorders) | 13 (13)
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 89 (89)
Hyperglycemia (Metabolism and nutrition disorders) | 79 (79)
Hyperkalemia (Metabolism and nutrition disorders) | 9 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 16 (16)
Hypocalcemia (Metabolism and nutrition disorders) | 41 (41)
Hypoglycemia (Metabolism and nutrition disorders) | 10 (10)
Hypokalemia (Metabolism and nutrition disorders) | 12 (12)
Hypomagnesemia (Metabolism and nutrition disorders) | 10 (10)
Hyponatremia (Metabolism and nutrition disorders) | 10 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 33 (33)
Infection without neutropenia (Infections and infestations) | 5 (5)
Leukocytes (Blood and lymphatic system disorders) | 68 (68)
Lymphopenia (Blood and lymphatic system disorders) | 94 (94)
Neutrophils (Blood and lymphatic system disorders) | 64 (64)
Platelets (Blood and lymphatic system disorders) | 70 (70)
Prothrombin time (PT) (Blood and lymphatic system disorders) | 9 (9)
Partial thromboplastin time (PTT) (Blood and lymphatic system disorders) | 15 (15)
SGOT (AST) (Blood and lymphatic system disorders) | 22 (22)
SGPT (ALT) (Blood and lymphatic system disorders) | 30 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes